CLINICAL TRIAL: NCT00746707
Title: Randomized Control Trial for the Comparison of Biologic Glue Versus Suturing for First Degree Perineal Tears
Brief Title: Biologic Glue for First Degree Perineal Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ezra Yosi, MD, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: feigenberg HMO-CTIL
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Grade 1 Perineal Tears
Keywords: adhesive glue, perineal tear, suture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): use of octyl-2-cyanoacrylate adhesive glue for perineal tear grade 1 in 80 women
  Interventions: Device: 1. Dermabond Topical Skin Adhesive 2-Octyl Cyanoacrylate
- 3 (Active Comparator): use of traditional suturing for perineal tear grade 1 in 50 women
  Interventions: Procedure: 3. traditional suturing with vicryl rapid 2X0

INTERVENTIONS:
Device: 1. Dermabond Topical Skin Adhesive 2-Octyl Cyanoacrylate — adhesive of perineal tears
  Arms: 1
Procedure: 3. traditional suturing with vicryl rapid 2X0 — suturing of perineal tears grade one with vicryl rapid 2X0
  Arms: 3

SUMMARY:
The use of octyl-2-cyanoacrylate adhesive glue is not inferior to traditional suturing for first degree perineal tears repair

DETAILED DESCRIPTION:
This is a prospective randomized trial, comparing the use of octyl-2-cyanoacrylate adhesive glue to traditional suturing, for the repair of first degree perineal tears.

ELIGIBILITY:
Inclusion Criteria:

* women after instrumental or normal vaginal delivery with a diagnosis of first degree perineal tears

Exclusion Criteria:

* excessive bleeding,
* chronic steroid treatment,
* immunosuppressive treatment,
* active infection,
* allergy to Dermabond or Histoacryl

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Functional and cosmetic evaluation of perineal tear area. | At least six weeks after birth

SECONDARY OUTCOMES:
Assessment of pain at least six weeks after delivery | At least six weeks after delivery

CONTACTS AND LOCATIONS:
Overall Officials: yosef ezra, M.D., Study Director — hadassha medical organization, jerusalem israel
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Feigenberg T, Maor-Sagie E, Zivi E, Abu-Dia M, Ben-Meir A, Sela HY, Ezra Y. Using adhesive glue to repair first degree perineal tears: a prospective randomized controlled trial. Biomed Res Int. 2014;2014:526590. doi: 10.1155/2014/526590. Epub 2014 Jun 26. PMID 25089271